CLINICAL TRIAL: NCT05260840
Title: Establishing and Evaluating a Beverage Intake Measurement Tool for the UK Workplace: The Fluid at Work Study
Brief Title: Fluid at Work Study
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: British Dietetic Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: GET2019
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: Workplace; Fluid; Assessment; Employee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — If participants consent, a urine sample will bio banked for future analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation study - provision of an online questionnaire — Evaluation study - provision of an online questionnaire

SUMMARY:
The aim of the Fluid at Work Study is to develop and evaluate a fluid intake measurement tool for use in the UK working population.

From the results of a systematic review and a round table discussion a novel fluid measurement tool has been developed - the Workplace Beverage Intake Questionnaire (WBIQ)

The observational evaluation study will measure the relative validity and reliability of WBIQ for assessing fluid intake in a workplace population.

DETAILED DESCRIPTION:
The aim of the Fluid at Work Study is to develop and evaluate a fluid intake measurement tool for use in the UK working population.

From the results of a systematic review and a round table discussion a novel fluid measurement tool has been developed - the Workplace Beverage Intake Questionnaire (WBIQ)

WBIQ will be used to conduct a preliminary investigation of relative validity and reliability. Relative validity of the tool will be tested, rather than 'absolute validity', as there is no 'gold' standard measure for exact fluid intake in free living population groups.

Individuals responding to local advertisements will complete an initial telephone or email questionnaire, and then eligible respondents will be asked to attend King's College London for a screening visit where they will be asked questions to confirm their inclusion criteria. Inclusion criteria: full-time disked based/ office workers. Following confirmation of eligibility and written consent participants will be asked to attend two study visits 7-days apart and complete three on-line fluid intake surveys.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employee working in a desk-based role
* No history of heart attack, stroke, angina, thrombosis, liver or kidney diseases, diabetes, chronic gastrointestinal disorder, or cancer
* Able to remain within the UK during the 8-10-week period of testing
* No history of excess alcohol intake or substance abuse
* Agree to not drink alcohol for the 7-day period of dietary data collection
* Not already participating in a clinical trial
* Not currently taking medication that is likely to alter kidney function or fluid balance
* Able to understand the information sheet and willing to comply with study protocol
* Able to give informed written consent

Exclusion Criteria:

* Pregnant or breast feeding

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Desk based office employees
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Relative validity of fluid intake measurement | 7 days
  Measured against 24-hr urine output, specific gravity and 7 day reported fluid intake
Reliability of fluid intake measurement (l/day) | 2 months
  Comparison of WBIQ responses at 3 time points

CONTACTS AND LOCATIONS:
Locations (1):
- Life Course Sciences, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided